CLINICAL TRIAL: NCT02956187
Title: Effect of Treatment of Constipation on Dyspeptic Symptoms in Patients With Constipation and Functional Dyspepsia
Brief Title: Treatment of Constipation in Functional Dyspepsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PR(AG)181/2016
Record Dates: First submitted 2016-08-04; First posted 2016-11-07 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2016-09

CONDITIONS: Dyspepsia; Constipation
MeSH Terms: conditions — Dyspepsia; Constipation | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biofeedback for constipation (Experimental): Constipation will be treated by correcting functional outlet obstruction.
  Interventions: Behavioral: Biofeedback
- Fiber supplementation (Active Comparator): Constipation will be treated by a fiber supplement
  Interventions: Dietary Supplement: Fiber supplement

INTERVENTIONS:
Behavioral: Biofeedback — Functional outlet obstruction will be treated by biofeedback: sessions of biofeedback guided by anorectal manometry combined with instructions for daily exercizing for 4 weeks.
  Arms: Biofeedback for constipation
Dietary Supplement: Fiber supplement — 3.5 g plantago ovata per day will be administered for 4 weeks.
  Arms: Fiber supplementation

SUMMARY:
Background. Functional dyspepsia is characterized by symptoms that apparently originate in the stomach without detectable cause by conventional diagnosis test. The pathophysiology of functional dyspepsia is not known, but a number of data indicate that dyspeptic patients have increased sensitivity of the digestive system, so that physiological stimuli may induce their symptoms. Some patients with functional dyspepsia have also functional constipation and the investigators hypothesize that in them constipation triggers or facilitates dyspeptic symptoms, and consequently, correction of constipation relieves dyspeptic symptoms.

Objective. To demonstrate the superiority of biofeedback versus a fiber supplement for the treatment of dyspeptic symptoms in patients with constipation due to functional outlet obstruction.

Design. Randomized, controlled parallel trial performed in a referral center. Participants. Consecutive patients complaining of symptoms of functional dyspepsia and functional outlet obstruction.

Interventions: Patients will be assigned to experimental (biofeedback for functional outlet obstruction) and active comparator (fiber supplementation) arms. Biofeedback for functional outlet obstruction: sessions of biofeedback guided by anorectal manometry (performed during the first 3 weeks of the intervention period) combined with instructions for daily exercising for 4 weeks. Fiber supplementation: 2.5 g plantago ovata per day for 4 weeks. Main outcome and measures. Clinical symptoms of functional dyspepsia measured by daily questionnaires for 7 consecutive days before and during the last week of intervention.

Relevance. Functional Dyspepsia, defined by purely clinical criteria, brings together a diverse group of conditions with different pathophysiology. As a result, the treatment is empirical and globally inefficient. This study will identify a subset of patients with a common pathophysiological mechanism of dyspeptic symptoms (functional outlet obstruction) which respond to specific treatment (biofeedback).

ELIGIBILITY:
Patients with functional dyspepsia and functional constipation.

Inclusion Criteria

* Rome IV criteria for functional dyspepsia type of postprandial distress syndrome.
* Rome IV criteria of functional constipation
* Anorectal manometry showing defective sphincter relaxation during the defecatory manoeuver.

Exclusion Criteria:

* History of organic gastrointestinal disorders
* Cognitive impairment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06-12; Primary Completion 2017-12-10 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
Change in clinical symptoms of functional dyspepsia during treatment versus before. | 4 weeks
  Change in average postprandial abdominal fullness measured daily by 0-10 score scales for 7 consecutive days before and during the last week of intervention.

SECONDARY OUTCOMES:
Change in postprandial abdominal fullness measured after a test meal by the end of treatment versus before | 4 weeks
  Change in average postprandial abdominal fullness measured by 0-10 score scales at the end of the test meal administered before and after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Azpiroz, MD, Principal Investigator — Principal Investigator
Locations (1):
- Fernando Azpiroz, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huaman JW, Mego M, Bendezu A, Monrroy H, Samino S, Accarino A, Saperas E, Azpiroz F. Correction of Dyssynergic Defecation, but Not Fiber Supplementation, Reduces Symptoms of Functional Dyspepsia in Patients With Constipation in a Randomized Trial. Clin Gastroenterol Hepatol. 2020 Oct;18(11):2463-2470.e1. doi: 10.1016/j.cgh.2019.11.048. Epub 2019 Dec 4. PMID 31811952